CLINICAL TRIAL: NCT01204658
Title: Safety, Reactogenicity & Immunogenicity of GSK Biologicals' Pneumococcal Vaccine 2189242A When Co-administered With DTPa-HBV-IPV/Hib Vaccine in Healthy Infants
Brief Title: Safety & Immunogenicity of Pneumococcal Vaccine 2189242A Co-administered With DTPa-HBV-IPV/Hib in Healthy Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 113994; 2010-019730-27 (EudraCT Number)
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Results first posted 2016-09-28 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Infections, Streptococcal
Keywords: Haemophilus influenzae; Streptococcus pneumoniae; immunogenicity; Pneumococcal vaccine; infants; safety
MeSH Terms: conditions — Streptococcal Infections; Haemophilus Infections | interventions — PHiD-CV vaccine; 13-valent pneumococcal vaccine; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 10PP-LD/Infanrix hexa Group (Experimental): This group consisted in infants aged 6-14 weeks at primary vaccination who received a 3-dose primary vaccination of the GSK 2189242A (or 10PP) vaccine combined with low doses (LD) of pneumococcal pneumolysin toxoid proteins (dPly) and pneumococcal histidine protein D (PhtD) co-administered with the Infanrix hexa™ vaccine at Study Months 0, 1 and 2. Subjects also received a booster dose of each of these vaccines, administered at Study Month 10. The 3 primary doses of the 10PP and Infanrix hexa™ vaccines were administered intramuscularly (IM) in the thigh, on the right and left side, respectively. Booster doses were administered IM into the deltoid or thigh if the deltoid muscle size was not adequate, on the left side for the 10PP vaccine and on the right side for Infanrix hexa™.
  Interventions: Biological: Pneumococcal vaccine GSK 2189242A (LD formulation 1); Biological: Infanrix Hexa (DTPa-HBV-IPV/Hib)
- 10PP-HD/Infanrix hexa Group (Experimental): This group consisted in infants aged 6-14 weeks at primary vaccination who received a 3-dose primary vaccination of the GSK 2189242A (or 10PP) vaccine combined with high doses (HD) of pneumococcal pneumolysin toxoid proteins (dPly) and pneumococcal histidine protein D (PhtD), co-administered with the Infanrix hexa™ vaccine at Study Months 0, 1 and 2. Subjects also received a booster dose of each of these vaccines, administered at Study Month 10. The 3 primary doses of the 10PP and Infanrix hexa™ vaccines were administered intramuscularly (IM) in the thigh, on the right and left side, respectively. Booster doses were administered IM into the deltoid or thigh if the deltoid muscle size was not adequate, on the left side for the 10PP vaccine and on the right side for Infanrix hexa™.
  Interventions: Biological: Pneumococcal vaccine GSK 2189242A (HD formulation 2); Biological: Infanrix Hexa (DTPa-HBV-IPV/Hib)
- Synflorix/Infanrix hexa Group (Active Comparator): This group consisted in infants aged 6-14 weeks at primary vaccination who received a 3-dose primary vaccination of Synflorix™ vaccine, co-administered with the Infanrix hexa™ vaccine at Study Months 0, 1 and 2. Subjects also received a booster dose of each of these vaccines, administered at Study Month 10. The 3 primary doses of Synflorix™ and Infanrix hexa™ vaccines were administered intramuscularly (IM) in the thigh, on the right and left side, respectively. Booster doses were administered IM into the deltoid or thigh if the deltoid muscle size was not adequate, on the left side for Synflorix™ and on the right side for Infanrix hexa™.
  Interventions: Biological: Synflorix; Biological: Infanrix Hexa (DTPa-HBV-IPV/Hib)
- Prevnar 13/Infanrix hexa Group (Active Comparator): This group consisted in infants aged 6-14 weeks at primary vaccination who received a 3-dose primary vaccination of Prevnar 13™ vaccine, co-administered with the Infanrix hexa™ vaccine at Study Months 0, 1 and 2. Subjects also received a booster dose of each of these vaccines, administered at Study Month 10. The 3 primary doses of Prevnar 13™ and Infanrix hexa™ vaccines were administered intramuscularly (IM) in the thigh, on the right and left side, respectively. Booster doses were administered IM into the deltoid or thigh if the deltoid muscle size was not adequate, on the left side for Prevnar 13™ and on the right side for Infanrix hexa™.
  Interventions: Biological: Prevenar 13; Biological: Infanrix Hexa (DTPa-HBV-IPV/Hib)

INTERVENTIONS:
Biological: Pneumococcal vaccine GSK 2189242A (LD formulation 1) — Intramuscular injection
  Other Names: GSK 2189242A; 10PP-LD
  Arms: 10PP-LD/Infanrix hexa Group
Biological: Pneumococcal vaccine GSK 2189242A (HD formulation 2) — Intramuscular injection
  Other Names: GSK 2189242A; 10PP-HD
  Arms: 10PP-HD/Infanrix hexa Group
Biological: Synflorix — Intramuscular injection
  Arms: Synflorix/Infanrix hexa Group
Biological: Prevenar 13 — Intramuscular injection
  Arms: Prevnar 13/Infanrix hexa Group
Biological: Infanrix Hexa (DTPa-HBV-IPV/Hib) — Intramuscular injection

SUMMARY:
This study will assess the safety, reactogenicity and immunogenicity of two formulations of GSK Biologicals' pneumococcal vaccine 2189242A given as a 3-dose primary vaccination course during the first 6 months of life followed by a booster dose at 12-15 months of age and co-administered with DTPa-HBV-IPV/Hib vaccine.

DETAILED DESCRIPTION:
This study will assess the safety, reactogenicity, immunogenicity and persistence of two formulations of GSK Biologicals' pneumococcal vaccine 2189242A [high dose (HD) or low dose (LD)] given as a 3-dose primary vaccination course during the first 6 months of life followed by a booster dose at 12-15 months of age when co-administered with Infanrix hexa™ and compared to the vaccination with Synflorix™ and with Prevnar 13™ similarly co-administered with the Infanrix hexa™ vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) (LAR) can and will comply with the requirements of the protocol
* Male or female between, and including, 6 and 14 weeks (42-104 days) of age at the time of the first vaccination.
* Written informed consent obtained from the parents/LAR(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born after a gestation period of 36 to 42 weeks inclusive.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/administration of a vaccine not foreseen by the study protocol during the study period starting from 30 days before each dose and ending 30 days after each dose of vaccine(s), with the exception of licensed flu vaccines.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Previous vaccination against S. pneumoniae since birth.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s).
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency.
* Major congenital defects or any chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease and/or fever at the time of enrolment.
* Fever is defined as temperature >= 38.0°C on rectal setting or >= 37.5°C on oral or axillary setting.
* Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/ or any blood products since birth or planned administration during the primary epoch and during the period starting three months before booster vaccination and ending one month after the booster vaccination.

Ages: 6 Weeks to 14 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 576 (Actual)
Dates: Start 2010-09-27 (Actual); Primary Completion 2011-11-03 (Actual); Study Completion 2012-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (24):
- Czechia (10):
  - GSK Investigational Site, Benešov
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Děčín
  - GSK Investigational Site, Jindřichův Hradec
  - GSK Investigational Site, Kladno
  - GSK Investigational Site, Liberec
  - GSK Investigational Site, Náchod
  - GSK Investigational Site, Ostrov
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Prague
- Germany (5):
  - GSK Investigational Site, Schwäbisch Hall, Baden-Wurttemberg
  - GSK Investigational Site, Tuttlingen, Baden-Wurttemberg
  - GSK Investigational Site, Detmold, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Berlin
- Poland (6):
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Sweden (3):
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Östersund
  - GSK Investigational Site, Umeå

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Prymula R, Szenborn L, Silfverdal SA, Wysocki J, Albrecht P, Traskine M, Gardev A, Song Y, Borys D. Safety, reactogenicity and immunogenicity of two investigational pneumococcal protein-based vaccines: Results from a randomized phase II study in infants. Vaccine. 2017 Aug 16;35(35 Pt B):4603-4611. doi: 10.1016/j.vaccine.2017.07.008. Epub 2017 Jul 17. PMID 28729019

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 576 subjects were initially enrolled in the study. Of these, one subject was older than protocol defined age range for the first vaccination, and therefore did not receive any vaccination.
Pre-assignment Details: The study duration is approximately 10 to 14 months depending on age at recruitment and age at booster vaccination. 2 Phases in the study: Primary Phase when subjects received a 3-dose of pneumococcal vaccine co-administered with Infanrix hexa™ (Months 0, 1, 2), and Booster Phase when subjects received one dose of the same vaccines (Month 10).
Period: Primary Phase
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Started | 146 | 142 | 145 | 142
Completed | 146 | 142 | 144 | 142
Not Completed | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: Booster Phase
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Started | 144 (Not all subjects completing the primary vaccination returned for the booster phase.) | 140 (Not all subjects completing the primary vaccination returned for the booster phase.) | 140 (Not all subjects completing the primary vaccination returned for the booster phase.) | 140 (Not all subjects completing the primary vaccination returned for the booster phase.)
Completed | 144 | 140 | 140 | 140
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group | Total
Number analyzed (Participants) | 146 | 142 | 145 | 142 | 575
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 10.3 (2.49) | 10.1 (2.70) | 10.1 (2.61) | 10.2 (2.64) | 10.2 (2.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 67 | 70 | 66 | 268
  Male | 81 | 75 | 75 | 76 | 307

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any and Grade 3 Solicited General Symptoms and With Solicited General Symptoms Related to Vaccination - Primary Phase of the Study
Description: Assessed solicited general symptoms were Drowsiness, Irritability, Loss of appetite (Loss Appet.) and Fever (rectal temperature higher than or equal to [>=] 38 degrees Celsius [°C]). Any = Occurrence of the specified solicited general symptom, regardless of intensity and relationship to vaccination. Related = Occurrence of the specified symptom assessed by the investigators as causally related to vaccination. Grade 3 (G3) Drowsiness = Drowsiness that prevented normal activity. G3 Irritability = Crying that could not be comforted/prevented normal activity. G3 Loss of appetite = Subject did not eat at all. G3 Fever = Rectal temperature higher than (>) 40.0°C. Primary results correspond to results for occurrences of G3 fever symptoms assessed by the investigators as related to vaccination (Related G3 fever).
Time Frame: Within the 7-day (Days 0-6) periods post vaccination, after each dose (D) of the 3-dose primary vaccination course
Population: The analysis was performed on the Total Vaccinated cohort for the Primary Phase, which included all subjects who received at least one of the 3 vaccine doses against pneumococcal diseases, with analysis done solely on subjects with post-vaccination solicited symptoms results available.
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 146 | 142 | 144 | 142
Participants
  Any Drowsiness, post D1 | 82 | 76 | 72 | 77
  G3 Drowsiness, post D1 | 4 | 0 | 2 | 2
  Related Drowsiness, post D1 | 63 | 58 | 52 | 58
  Any Irritability, post D1 | 93 | 82 | 89 | 82
  G3 Irritability, post D1 | 6 | 9 | 9 | 5
  Related Irritability, post D1 | 70 | 62 | 66 | 57
  Any Loss Appet., post D1 | 38 | 32 | 39 | 32
  G3 Loss Appet., post D1 | 0 | 1 | 0 | 0
  Related Loss Appet., post D1 | 28 | 26 | 29 | 21
  Any Fever, post D1 | 45 | 32 | 53 | 28
  G3 Fever, post D1 | 0 | 0 | 0 | 0
  Related Fever, post D1 | 33 | 25 | 44 | 27
  Related G3 Fever, post D1 | 0 | 0 | 0 | 0
  Any Drowsiness, post D2 | 71 | 63 | 70 | 66
  G3 Drowsiness, post D2 | 4 | 2 | 1 | 1
  Related Drowsiness, post D2 | 53 | 49 | 56 | 55
  Any Irritability, post D2 | 88 | 81 | 86 | 87
  G3 Irritability, post D2 | 8 | 3 | 5 | 6
  Related Irritability, post D2 | 69 | 66 | 66 | 67
  Any Loss Appet., post D2 | 32 | 30 | 28 | 30
  G3 Loss Appet., post D2 | 1 | 2 | 0 | 0
  Related Loss Appet., post D2 | 23 | 21 | 18 | 25
  Any Fever, post D2 | 40 | 50 | 38 | 38
  G3 Fever, post D2 | 0 | 0 | 0 | 0
  Related Fever, post D2 | 32 | 39 | 33 | 31
  Related G3 Fever, post D2 | 0 | 0 | 0 | 0
  Any Drowsiness, post D3: number analyzed (Participants) | 146 | 141 | 143 | 142
  Any Drowsiness, post D3 | 57 | 48 | 56 | 48
  Grade 3 Drowsiness, post D3: number analyzed (Participants) | 146 | 141 | 143 | 142
  Grade 3 Drowsiness, post D3 | 2 | 0 | 1 | 1
  Related Drowsiness, post D3: number analyzed (Participants) | 146 | 141 | 143 | 142
  Related Drowsiness, post D3 | 51 | 38 | 44 | 36
  Any Irritability, post D3: number analyzed (Participants) | 146 | 141 | 143 | 142
  Any Irritability, post D3 | 62 | 73 | 62 | 72
  G3 Irritability, post D3: number analyzed (Participants) | 146 | 141 | 143 | 142
  G3 Irritability, post D3 | 7 | 1 | 3 | 2
  Related Irritability, post D3: number analyzed (Participants) | 146 | 141 | 143 | 142
  Related Irritability, post D3 | 52 | 55 | 48 | 53
  Any Loss Appet., post D3: number analyzed (Participants) | 146 | 141 | 143 | 142
  Any Loss Appet., post D3 | 28 | 25 | 24 | 21
  G3 Loss Appet., post D3: number analyzed (Participants) | 146 | 141 | 143 | 142
  G3 Loss Appet., post D3 | 0 | 0 | 2 | 2
  Related Loss Appet., post D3: number analyzed (Participants) | 146 | 141 | 143 | 142
  Related Loss Appet., post D3 | 22 | 20 | 18 | 13
  Any Fever, post D3: number analyzed (Participants) | 146 | 141 | 143 | 142
  Any Fever, post D3 | 28 | 23 | 27 | 30
  G3 Fever, post D3: number analyzed (Participants) | 146 | 141 | 143 | 142
  G3 Fever, post D3 | 0 | 0 | 0 | 0
  Related Fever, post D3: number analyzed (Participants) | 146 | 141 | 143 | 142
  Related Fever, post D3 | 23 | 19 | 20 | 22
  Related G3 Fever, post D3: number analyzed (Participants) | 146 | 141 | 143 | 142
  Related G3 Fever, post D3 | 0 | 0 | 0 | 0

2. Primary Outcome: Percentage of Subjects Reporting Fever > 40.0°C With Causal Relationship to Vaccination After Each Primary Vaccination Dose and Across Doses in 10PP-LD/Infanrix Hexa Group and in Synflorix/Infanrix Hexa Group
Description: Grade 3 fever was defined as fever by rectal measurement > 40.0°C. Related was defined as causal relationship to vaccination. This endpoint was assessed after each primary vaccination dose and across doses and in subjects in the 10PP-LD/Infanrix hexa (or 10PP-LD) and Synflorix/Infanrix hexa (or 10PN) groups only.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each primary vaccination dose and across doses
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 10PP-LD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group
Number analyzed (Participants) | 146 | 144
Percentage of participants
  Fever>40.0°C & Related Dose 1 | 0.0 | 0.0
  Fever>40.0°C & Related Dose 2 | 0.0 | 0.0
  Fever>40.0°C & Related Dose 3: number analyzed (Participants) | 146 | 143
  Fever>40.0°C & Related Dose 3 | 0.0 | 0.0
  Fever>40.0°C & Related across doses | 0.0 | 0.0
Statistical Analysis 1: Comparison: 10PP-LD/Infanrix Hexa Group vs Synflorix/Infanrix Hexa Group; Non-inferiority of 10PP-LD vaccine vs Synflorix™ vaccine post dose 1 was assessed by computing the difference in percentages of subjects reporting Grade 3 fever causally related to dose 1 vaccination in the 10PP-LD Group minus Synflorix Group; Test type: Non-Inferiority or Equivalence — Non-inferiority was supported if one could rule out an increase in terms of percentage of subjects (10PP-LD Group minus Synflorix Group) above 5% + half the incidence in the Synflorix Group (= null hypothesis) as shown by a 1-sided P-value < 5%; p = 0.003, Kem Phillip's statistical test — 1-sided P-value computed using Kem Philips' approach for ruling out an increase in % subjects with fever > 40.0°C and causal relationship to vaccination > the boundary expressed as 5% + 0.5*rate in the Synflorix group; Difference in percentage = 0, 95% CI 2-sided [-2.61 to 2.57]
Statistical Analysis 2: Comparison: 10PP-LD/Infanrix Hexa Group vs Synflorix/Infanrix Hexa Group; Non-inferiority of 10PP-LD vaccine vs Synflorix™ vaccine post dose 2 was assessed by computing the difference in percentages of subjects reporting Grade 3 fever causally related to dose 2 vaccination in the 10PP-LD Group minus Synflorix Group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.003, Kem Phillip's statistical test — [p-value comment as in outcome 2, analysis 1]; Difference in percentage = 0, 95% CI 2-sided [-2.61 to 2.57]
Statistical Analysis 3: Comparison: 10PP-LD/Infanrix Hexa Group vs Synflorix/Infanrix Hexa Group; Non-inferiority of 10PP-LD vaccine vs Synflorix™ vaccine post dose 3 was assessed by computing the difference in percentages of subjects reporting Grade 3 fever causally related to dose 3 vaccination in the 10PP-LD Group minus Synflorix Group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.003, Kem Phillip's statistical test — [p-value comment as in outcome 2, analysis 1]; Difference in percentage = 0, 95% CI 2-sided [-2.62 to 2.57]
Statistical Analysis 4: Comparison: 10PP-LD/Infanrix Hexa Group vs Synflorix/Infanrix Hexa Group; Non-inferiority of 10PP-LD vaccine vs Synflorix™ vaccine across doses was assessed by computing the difference in percentages of subjects reporting Grade 3 fever causally related to vaccination, across doses, in the 10PP-LD Group minus Synflorix Group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.003, Kem Phillip's statistical test — [p-value comment as in outcome 2, analysis 1]; Difference in percentage = 0, 95% CI 2-sided [-2.61 to 2.57]

3. Primary Outcome: Percentage of Subjects Reporting Fever > 40° C With Causal Relationship to Vaccination After Each Primary Vaccination Dose and Across Doses in the 10PP-HD/Infanrix Hexa Group and in the Synflorix/Infanrix Hexa Group
Description: Grade 3 fever was defined as fever by rectal measurement >40.0°C. Related was defined as causal relationship to vaccination. This endpoint was assessed after each primary vaccination dose and across doses and in subjects in the 10PP-HD/Infanrix hexa (or 10PP-HD) and Synflorix/Infanrix hexa (or 10PN) groups only.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each primary vaccination dose and across doses
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group
Number analyzed (Participants) | 142 | 144
Percentage of participants
  Fever>40.0°C & Related Dose 1 | 0.0 | 0.0
  Fever>40.0°C & Related Dose 2 | 0.0 | 0.0
  Fever>40.0°C & Related Dose 3: number analyzed (Participants) | 141 | 143
  Fever>40.0°C & Related Dose 3 | 0.0 | 0.0
  Fever>40.0°C & Related across doses | 0.0 | 0.0
Statistical Analysis 1: Comparison: 10PP-HD/Infanrix Hexa Group vs Synflorix/Infanrix Hexa Group; Non-inferiority of 10PP-HD vaccine vs Synflorix™ vaccine post dose 1 was assessed by computing the difference in percentages of subjects reporting Grade 3 fever causally related to dose 1 vaccination in the 10PP-HD Group minus Synflorix Group; Test type: Non-Inferiority or Equivalence — Non-inferiority was supported if one could rule out an increase in terms of percentage of subjects (10PP-HD Group minus Synflorix Group) above 5% + half the incidence in the Synflorix Group (= null hypothesis) as shown by a 1-sided P-value < 5%; p = 0.003, Kem Phillip's statistical test — [p-value comment as in outcome 2, analysis 1]; Difference in percentage = 0, 95% CI 2-sided [-2.61 to 2.64]
Statistical Analysis 2: Comparison: 10PP-HD/Infanrix Hexa Group vs Synflorix/Infanrix Hexa Group; Non-inferiority of 10PP-HD vaccine vs Synflorix™ vaccine post dose 2 was assessed by computing the difference in percentages of subjects reporting Grade 3 fever causally related to dose 2 vaccination in the 10PP-HD Group minus Synflorix Group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.003, Kem Phillip's statistical test — [p-value comment as in outcome 2, analysis 1]; Difference in percentage = 0, 95% CI 2-sided [-2.61 to 2.64]
Statistical Analysis 3: Comparison: 10PP-HD/Infanrix Hexa Group vs Synflorix/Infanrix Hexa Group; Non-inferiority of 10PP-HD vaccine vs Synflorix™ vaccine post dose 3 was assessed by computing the difference in percentages of subjects reporting Grade 3 fever causally related to dose 3 vaccination in the 10PP-HD Group minus Synflorix Group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.003, Kem Phillip's statistical test — [p-value comment as in outcome 2, analysis 1]; Difference in percentage = 0, 95% CI 2-sided [-2.63 to 2.66]
Statistical Analysis 4: Comparison: 10PP-HD/Infanrix Hexa Group vs Synflorix/Infanrix Hexa Group; Non-inferiority of 10PP-HD vaccine vs Synflorix™ vaccine across doses was assessed by computing the difference in percentages of subjects reporting Grade 3 fever causally related to vaccination, across doses, in the 10PP-HD Group minus Synflorix Group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; p = 0.003, Kem Phillip's statistical test — [p-value comment as in outcome 2, analysis 1]; Difference in percentage = 0, 95% CI 2-sided [-2.61 to 2.64]

4. Secondary Outcome: Antibody Concentrations Against Pneumococcal Pneumolysin Toxoid (dPly) and Pneumococcal Histidine Triad Protein D (PhtD) Proteins - Primary Phase of the Study
Description: Antibody concentrations against dPly and PhtD (anti-dPly and anti-PhtD, respectively) were measured by enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in ELISA Units per milliliter (EL.U/mL). Cut-offs for seropositivity were concentrations higher than or equal to (≥)12 EL.U/mL for anti-dPly antibodies and ≥ 17 EL.U/mL for anti-PhtD antibodies. This outcome concerns results for the Primary Phase of the study.
Time Frame: At Month 3, e. g. one month post-Dose 3 of pneumococcal vaccine (10PP, Synflorix™ or Prevnar 13™)
Population: The analysis was performed on the According-To-Protocol cohort for immunogenicity adapted for each epoch which included all evaluable subjects for whom immunogenicity data were available for antibodies against at least one study antigen component after primary vaccination (primary phase) or before or after booster vaccination (booster phase).
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 130 | 134 | 136 | 131
EL.U/mL
  Anti-dPly - At Month 3 | 9408.42 [8182.15 to 10818.47] | 12137.96 [10641.83 to 13844.44] | 459.97 [398.31 to 531.18] | 472.88 [404.48 to 552.86]
  Anti-PhtD - At Month 3 | 1456.57 [1250.65 to 1696.39] | 1996.61 [1734.17 to 2298.75] | 523.61 [453.71 to 604.28] | 552.01 [469.55 to 648.95]

5. Secondary Outcome: Antibody Concentrations Against Pneumococcal Pneumolysin Toxoid (dPly) and Pneumococcal Histidine Triad Protein D (PhtD) Proteins - Booster Phase of the Study
Description: Antibody concentrations against dPly and PhtD (anti-dPly and anti-PhtD, respectively) were measured by enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in ELISA Units per milliliter (EL.U/mL). Cut-offs for seropositivity were concentrations higher than or equal to (≥)12 EL.U/mL for anti-dPly antibodies and ≥ 17 EL.U/mL for anti-PhtD antibodies. This outcome concerns results for the Booster Phase of the study.
Time Frame: At Months 10 and 11, e.g. prior to and at one month post booster vaccination with pneumococcal vaccine (10PP, Synflorix™ or Prevnar 13™)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 130 | 129 | 129 | 129
EL.U/mL
  Anti-dPly - Month 10: number analyzed (Participants) | 130 | 128 | 129 | 129
  Anti-dPly - Month 10 | 6674.42 [5628.57 to 7914.60] | 5592.85 [4750.83 to 6584.10] | 495.02 [393.19 to 623.22] | 737.71 [587.67 to 926.06]
  Anti-dPly - Month 11: number analyzed (Participants) | 129 | 129 | 129 | 125
  Anti-dPly - Month 11 | 24720.40 [21863.04 to 27951.19] | 29838.18 [26892.53 to 33106.48] | 582.85 [463.40 to 733.09] | 791.42 [628.23 to 997.00]
  Anti-PhtD - Month 10: number analyzed (Participants) | 130 | 128 | 129 | 129
  Anti-PhtD - Month 10 | 910.80 [718.85 to 1154.00] | 829.12 [671.12 to 1024.32] | 209.27 [153.16 to 285.95] | 381.66 [274.64 to 530.39]
  Anti-PhtD - Month 11: number analyzed (Participants) | 129 | 129 | 129 | 125
  Anti-PhtD - Month 11 | 3528.25 [2952.68 to 4216.01] | 3777.39 [3181.74 to 4484.55] | 266.58 [190.06 to 373.91] | 469.16 [335.29 to 656.46]

6. Secondary Outcome: Antibody Concentrations Against Protein D (Anti-PD) - Primary Phase of the Study
Description: Antibody concentrations were measured by enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in ELISA Units per milliliter (EL.U/mL). The seropositivity cut-off of the assay was a concentration of anti-PD antibodies ≥ 100 EL.U/mL. This outcome concerns results for the Primary Phase of the study.
Time Frame: At Month 3, e. g. one month post-Dose 3 of pneumococcal vaccine (10PP, Synflorix™ or Prevnar 13™)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 132 | 134 | 137 | 132
EL.U/mL | 1135.7 [927.8 to 1390.1] | 1323.3 [1099.7 to 1592.4] | 1539.0 [1258.4 to 1882.1] | 147.0 [112.3 to 192.3]

7. Secondary Outcome: Antibody Concentrations Against Protein D (Anti-PD) - Booster Phase of the Study
Description: Antibody concentrations were measured by enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in ELISA Units per milliliter (EL.U/mL). The seropositivity cut-off of the assay was a concentration of anti-PD antibodies ≥ 100 EL.U/mL. This outcome concerns results for the Booster Phase of the study.
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 131 | 130 | 131 | 129
EL.U/mL
  Anti-PD - Month 10 | 434.3 [365.5 to 516.0] | 472.8 [403.1 to 554.5] | 698.2 [593.7 to 821.0] | 81.0 [69.8 to 93.9]
  Anti-PD - Month 11: number analyzed (Participants) | 128 | 130 | 131 | 127
  Anti-PD - Month 11 | 1655.4 [1398.2 to 1960.0] | 1631.0 [1404.5 to 1894.2] | 2394.2 [2045.7 to 2802.1] | 85.7 [73.6 to 99.8]

8. Secondary Outcome: Antibody Concentrations Against Pneumococcal Serotypes - Primary Phase of the Study
Description: Antibodies assessed for this outcome measure were those against the vaccine/cross-reactive pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F (ANTI-1, -3, -4, -5, -6A, -6B, -7F, -9V, -14, -18C, -19A, -19F and -23F). Antibody concentrations were measured by 22F enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). The seropositivity cut-off of the assay was an antibody concentration ≥ 0.05 µg/mL. This outcome concerns results for the Primary Phase of the study.
Time Frame: At Month 3, e. g. one month post-Dose 3 of pneumococcal vaccine (10PP, Synflorix™ or Prevnar 13™)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 132 | 135 | 137 | 132
µg/mL
  ANTI-1 At Month 3: number analyzed (Participants) | 131 | 131 | 134 | 132
  ANTI-1 At Month 3 | 1.57 [1.36 to 1.80] | 1.58 [1.36 to 1.83] | 1.49 [1.28 to 1.74] | 2.20 [1.86 to 2.60]
  ANTI-4 At Month 3: number analyzed (Participants) | 131 | 133 | 133 | 132
  ANTI-4 At Month 3 | 2.04 [1.74 to 2.39] | 2.11 [1.83 to 2.43] | 1.82 [1.55 to 2.14] | 2.43 [2.05 to 2.88]
  ANTI-5 At Month 3: number analyzed (Participants) | 132 | 134 | 134 | 132
  ANTI-5 At Month 3 | 2.46 [2.13 to 2.85] | 2.55 [2.22 to 2.92] | 2.31 [2.00 to 2.67] | 2.77 [2.27 to 3.38]
  ANTI-6B At Month 3: number analyzed (Participants) | 130 | 129 | 133 | 132
  ANTI-6B At Month 3 | 0.36 [0.29 to 0.46] | 0.37 [0.31 to 0.45] | 0.40 [0.32 to 0.51] | 0.46 [0.37 to 0.57]
  ANTI-7F At Month 3: number analyzed (Participants) | 130 | 131 | 134 | 132
  ANTI-7F At Month 3 | 2.12 [1.86 to 2.41] | 2.21 [1.97 to 2.48] | 2.20 [1.92 to 2.50] | 2.94 [2.51 to 3.46]
  ANTI-9V At Month 3 | 1.83 [1.59 to 2.12] | 1.95 [1.73 to 2.20] | 1.99 [1.72 to 2.30] | 2.33 [1.96 to 2.76]
  ANTI-14 At Month 3: number analyzed (Participants) | 132 | 133 | 135 | 132
  ANTI-14 At Month 3 | 3.57 [3.08 to 4.14] | 3.72 [3.30 to 4.18] | 3.91 [3.41 to 4.48] | 4.18 [3.41 to 5.13]
  ANTI-18C At Month 3: number analyzed (Participants) | 132 | 132 | 135 | 132
  ANTI-18C At Month 3 | 2.27 [1.93 to 2.67] | 2.18 [1.84 to 2.59] | 2.45 [2.04 to 2.95] | 2.56 [2.14 to 3.07]
  ANTI-19F At Month 3: number analyzed (Participants) | 132 | 132 | 135 | 132
  ANTI-19F At Month 3 | 4.29 [3.63 to 5.07] | 4.13 [3.52 to 4.85] | 4.51 [3.79 to 5.36] | 3.50 [2.94 to 4.18]
  ANTI-23F At Month 3: number analyzed (Participants) | 131 | 133 | 135 | 132
  ANTI-23F At Month 3 | 0.67 [0.54 to 0.82] | 0.62 [0.50 to 0.78] | 0.67 [0.54 to 0.82] | 1.48 [1.17 to 1.88]
  ANTI-3 (At Month 3: number analyzed (Participants) | 130 | 129 | 132 | 132
  ANTI-3 (At Month 3 | 0.05 [0.04 to 0.06] | 0.06 [0.05 to 0.07] | 0.05 [0.05 to 0.06] | 2.47 [2.08 to 2.93]
  ANTI-6A At Month 3: number analyzed (Participants) | 129 | 132 | 133 | 132
  ANTI-6A At Month 3 | 0.13 [0.10 to 0.16] | 0.11 [0.09 to 0.14] | 0.11 [0.09 to 0.14] | 2.05 [1.69 to 2.50]
  ANTI-19A At Month 3: number analyzed (Participants) | 130 | 129 | 134 | 132
  ANTI-19A At Month 3 | 0.18 [0.14 to 0.23] | 0.17 [0.13 to 0.21] | 0.16 [0.13 to 0.20] | 2.77 [2.34 to 3.28]

9. Secondary Outcome: Antibody Concentrations Against Pneumococcal Serotypes - Booster Phase of the Study
Description: Antibodies assessed for this outcome measure were those against the vaccine/cross-reactive pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F (ANTI-1, -3, -4, -5, -6A, -6B, -7F, -9V, -14, -18C, -19A, -19F and -23F). Antibody concentrations were measured by 22F enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). The seropositivity cut-off of the assay was an antibody concentration higher than or equal to (≥) 0.05 µg/mL. This outcome concerns results for the Booster Phase of the study.
Time Frame: as for outcome 5
Population: The analysis was performed on the According-To-Protocol cohort for immunogenicity adapted for each epoch which included all evaluable subjects for whom immunogenicity data were available for antibodies against at least one study vaccine component after primary vaccination (primary phase) or before or after booster vaccination (booster phase).
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 130 | 131 | 131 | 129
µg/mL
  ANTI-1 Month 10: number analyzed (Participants) | 126 | 124 | 130 | 129
  ANTI-1 Month 10 | 0.30 [0.25 to 0.35] | 0.30 [0.26 to 0.36] | 0.26 [0.22 to 0.31] | 0.49 [0.43 to 0.55]
  ANTI-1 Month 11: number analyzed (Participants) | 130 | 131 | 131 | 127
  ANTI-1 Month 11 | 2.62 [2.27 to 3.04] | 2.61 [2.27 to 3.00] | 2.41 [2.06 to 2.82] | 3.78 [3.34 to 4.28]
  ANTI-4 Month 10: number analyzed (Participants) | 125 | 121 | 126 | 128
  ANTI-4 Month 10 | 0.50 [0.43 to 0.58] | 0.51 [0.43 to 0.61] | 0.58 [0.49 to 0.70] | 0.40 [0.35 to 0.46]
  ANTI-4 Month 11: number analyzed (Participants) | 130 | 129 | 131 | 127
  ANTI-4 Month 11 | 4.10 [3.54 to 4.74] | 3.90 [3.35 to 4.53] | 3.98 [3.51 to 4.52] | 4.36 [3.77 to 5.05]
  ANTI-5 Month 10: number analyzed (Participants) | 128 | 123 | 128 | 129
  ANTI-5 Month 10 | 0.59 [0.50 to 0.69] | 0.58 [0.49 to 0.68] | 0.55 [0.47 to 0.65] | 0.85 [0.74 to 0.99]
  ANTI-5 Month 11: number analyzed (Participants) | 129 | 129 | 131 | 127
  ANTI-5 Month 11 | 3.48 [2.98 to 4.05] | 3.44 [2.98 to 3.96] | 3.33 [2.87 to 3.87] | 7.52 [6.52 to 8.68]
  ANTI-6B Month 10: number analyzed (Participants) | 126 | 125 | 126 | 129
  ANTI-6B Month 10 | 0.45 [0.38 to 0.53] | 0.47 [0.39 to 0.56] | 0.46 [0.38 to 0.55] | 0.25 [0.21 to 0.31]
  ANTI-6B Month 11: number analyzed (Participants) | 129 | 129 | 131 | 127
  ANTI-6B Month 11 | 2.04 [1.77 to 2.36] | 1.96 [1.67 to 2.30] | 2.28 [1.94 to 2.68] | 3.11 [2.65 to 3.64]
  ANTI-7F Month 10: number analyzed (Participants) | 127 | 126 | 127 | 129
  ANTI-7F Month 10 | 0.94 [0.82 to 1.09] | 1.00 [0.88 to 1.15] | 0.98 [0.85 to 1.13] | 1.34 [1.18 to 1.53]
  ANTI-7F Month 11: number analyzed (Participants) | 129 | 129 | 131 | 127
  ANTI-7F Month 11 | 4.72 [4.13 to 5.40] | 4.70 [4.19 to 5.27] | 4.87 [4.32 to 5.50] | 7.68 [6.84 to 8.61]
  ANTI-9V Month 10: number analyzed (Participants) | 127 | 126 | 128 | 128
  ANTI-9V Month 10 | 0.77 [0.65 to 0.90] | 0.97 [0.84 to 1.12] | 0.99 [0.85 to 1.16] | 0.58 [0.50 to 0.68]
  ANTI-9V Month 11: number analyzed (Participants) | 129 | 129 | 131 | 127
  ANTI-9V Month 11 | 4.48 [3.90 to 5.14] | 4.91 [4.32 to 5.58] | 5.20 [4.52 to 5.97] | 6.57 [5.67 to 7.60]
  ANTI-14 Month 10: number analyzed (Participants) | 129 | 126 | 128 | 129
  ANTI-14 Month 10 | 1.36 [1.12 to 1.65] | 1.43 [1.18 to 1.73] | 1.57 [1.28 to 1.93] | 2.06 [1.72 to 2.47]
  ANTI-14 Month 11: number analyzed (Participants) | 129 | 129 | 131 | 127
  ANTI-14 Month 11 | 6.06 [5.18 to 7.09] | 7.18 [6.14 to 8.39] | 6.63 [5.59 to 7.86] | 11.43 [9.81 to 13.30]
  ANTI-18C Month 10: number analyzed (Participants) | 126 | 124 | 126 | 129
  ANTI-18C Month 10 | 0.75 [0.64 to 0.87] | 0.76 [0.65 to 0.89] | 0.92 [0.77 to 1.10] | 0.75 [0.65 to 0.85]
  ANTI-18C Month 11: number analyzed (Participants) | 129 | 129 | 131 | 127
  ANTI-18C Month 11 | 6.68 [5.76 to 7.75] | 6.38 [5.48 to 7.42] | 7.65 [6.76 to 8.67] | 6.40 [5.50 to 7.45]
  ANTI-19F Month 10: number analyzed (Participants) | 127 | 126 | 127 | 128
  ANTI-19F Month 10 | 1.25 [1.05 to 1.47] | 1.13 [0.96 to 1.33] | 1.30 [1.06 to 1.58] | 0.66 [0.53 to 0.82]
  ANTI-19F Month 11: number analyzed (Participants) | 130 | 129 | 131 | 127
  ANTI-19F Month 11 | 6.73 [5.77 to 7.83] | 7.22 [6.25 to 8.33] | 7.84 [6.78 to 9.06] | 7.43 [6.35 to 8.69]
  ANTI-23F Month 10: number analyzed (Participants) | 126 | 123 | 125 | 128
  ANTI-23F Month 10 | 0.46 [0.38 to 0.56] | 0.47 [0.38 to 0.58] | 0.57 [0.48 to 0.68] | 0.37 [0.30 to 0.44]
  ANTI-23F Month 11: number analyzed (Participants) | 129 | 129 | 131 | 127
  ANTI-23F Month 11 | 3.20 [2.68 to 3.83] | 3.20 [2.70 to 3.78] | 3.72 [3.21 to 4.31] | 7.10 [6.05 to 8.35]
  ANTI-3 Month 10: number analyzed (Participants) | 125 | 126 | 129 | 128
  ANTI-3 Month 10 | 0.05 [0.04 to 0.06] | 0.05 [0.04 to 0.06] | 0.05 [0.04 to 0.06] | 0.32 [0.27 to 0.38]
  ANTI-3 Month 11: number analyzed (Participants) | 128 | 128 | 131 | 127
  ANTI-3 Month 11 | 0.06 [0.05 to 0.08] | 0.05 [0.04 to 0.07] | 0.06 [0.05 to 0.07] | 1.83 [1.58 to 2.12]
  ANTI-6A Month 10: number analyzed (Participants) | 129 | 127 | 128 | 129
  ANTI-6A Month 10 | 0.19 [0.15 to 0.24] | 0.18 [0.15 to 0.22] | 0.20 [0.16 to 0.24] | 0.70 [0.59 to 0.83]
  ANTI-6A Month 11: number analyzed (Participants) | 130 | 130 | 131 | 127
  ANTI-6A Month 11 | 0.89 [0.72 to 1.11] | 0.74 [0.59 to 0.93] | 0.99 [0.78 to 1.26] | 7.77 [6.60 to 9.14]
  ANTI-19A Month 10: number analyzed (Participants) | 126 | 124 | 128 | 129
  ANTI-19A Month 10 | 0.18 [0.15 to 0.22] | 0.15 [0.12 to 0.18] | 0.18 [0.14 to 0.22] | 0.57 [0.44 to 0.73]
  ANTI-19A Month 11: number analyzed (Participants) | 128 | 128 | 131 | 127
  ANTI-19A Month 11 | 1.12 [0.89 to 1.41] | 1.03 [0.80 to 1.31] | 1.23 [0.99 to 1.52] | 7.77 [6.43 to 9.39]

10. Secondary Outcome: Titers for Opsonophagocytic Activity Against Pneumococcal Serotypes - Primary Phase of the Study
Description: Titers for opsonophagocytic activity assessed for this outcome measure were those for opsonophagocytic activity against the vaccine/cross-reactive pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F (OPA-1, -3, -4, -5, -6A, -6B, -7F, -9V, -14, -18C, -19A, -19F and -23F). The Seropositivity cut-off of the assay was a titer for opsonophagocytic activity higher than or equal to (≥) 8, except for the OPA-19A for which the titer was ≥ to the serotype-specific Lower Limit of Quantification (=143). This outcome concerns results for the Primary Phase of the study.
Time Frame: At Month 3, e. g. one month post-Dose 3 of pneumococcal vaccine (10PP, Synflorix™ or Prevnar 13™)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 63 | 57 | 66 | 63
Titers
  OPA-1 At Month 3: number analyzed (Participants) | 63 | 57 | 65 | 62
  OPA-1 At Month 3 | 38.6 [24.6 to 60.5] | 27.8 [17.5 to 44.2] | 29.4 [19.4 to 44.5] | 68.9 [47.5 to 99.9]
  OPA-4 At Month 3: number analyzed (Participants) | 60 | 57 | 66 | 63
  OPA-4 At Month 3 | 703.7 [533.5 to 928.2] | 844.4 [660.8 to 1079.0] | 819.2 [652.7 to 1028.1] | 748.1 [509.9 to 1097.5]
  OPA-5 At Month 3: number analyzed (Participants) | 63 | 56 | 65 | 63
  OPA-5 At Month 3 | 47.3 [33.6 to 66.6] | 60.6 [44.1 to 83.3] | 50.3 [37.2 to 68.1] | 72.9 [52.2 to 101.8]
  OPA-6B At Month 3: number analyzed (Participants) | 61 | 57 | 63 | 63
  OPA-6B At Month 3 | 399.6 [249.4 to 640.4] | 454.7 [299.8 to 689.7] | 409.7 [251.0 to 668.7] | 884.9 [569.3 to 1375.5]
  OPA-7F At Month 3: number analyzed (Participants) | 61 | 55 | 64 | 62
  OPA-7F At Month 3 | 3212.6 [2434.8 to 4238.8] | 3697.6 [2748.6 to 4974.1] | 4234.2 [3203.0 to 5597.4] | 7394.5 [4411.1 to 12395.7]
  OPA-9V At Month 3: number analyzed (Participants) | 60 | 56 | 64 | 62
  OPA-9V At Month 3 | 1942.4 [1381.9 to 2730.1] | 1520.7 [1109.4 to 2084.5] | 1983.6 [1507.2 to 2610.7] | 2242.8 [1474.7 to 3411.1]
  OPA-14 At Month 3: number analyzed (Participants) | 59 | 56 | 62 | 61
  OPA-14 At Month 3 | 1405.3 [1060.3 to 1862.4] | 1334.9 [1013.9 to 1757.4] | 1575.3 [1143.5 to 2170.1] | 2410.6 [1516.6 to 3831.5]
  OPA-18C At Month 3: number analyzed (Participants) | 58 | 52 | 59 | 58
  OPA-18C At Month 3 | 108.1 [72.6 to 161.2] | 102.7 [70.3 to 150.0] | 169.4 [121.9 to 235.4] | 257.6 [179.4 to 369.9]
  OPA-19F At Month 3: number analyzed (Participants) | 61 | 56 | 64 | 63
  OPA-19F At Month 3 | 211.6 [139.6 to 320.7] | 344.1 [240.6 to 492.0] | 381.6 [256.8 to 566.9] | 142.5 [98.9 to 205.4]
  OPA-23F At Month 3: number analyzed (Participants) | 60 | 54 | 63 | 63
  OPA-23F At Month 3 | 1275.6 [771.1 to 2110.3] | 2170.3 [1559.9 to 3019.6] | 1757.9 [1191.4 to 2593.7] | 4437.1 [2874.9 to 6848.2]
  OPA-3 (At Month 3: number analyzed (Participants) | 55 | 51 | 58 | 61
  OPA-3 (At Month 3 | 5.0 [3.9 to 6.4] | 4.5 [3.9 to 5.2] | 4.6 [4.0 to 5.3] | 88.4 [67.3 to 116.0]
  OPA-6A At Month 3: number analyzed (Participants) | 63 | 56 | 64 | 62
  OPA-6A At Month 3 | 43.2 [23.8 to 78.5] | 59.6 [35.4 to 100.3] | 44.7 [26.2 to 76.2] | 1726.0 [1113.9 to 2674.4]
  OPA-19A At Month 3: number analyzed (Participants) | 33 | 34 | 36 | 49
  OPA-19A At Month 3 | 576.0 [340.6 to 974.3] | 914.6 [586.8 to 1425.6] | 905.2 [628.2 to 1304.5] | 2915.3 [2270.3 to 3743.6]

11. Secondary Outcome: Titers for Opsonophagocytic Activity Against Pneumococcal Serotypes - Booster Phase of the Study
Description: Titers for opsonophagocytic activity assessed for this outcome measure were those for opsonophagocytic activity against the vaccine/cross-reactive pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F (OPA-1, -3, -4, -5, -6A, -6B, -7F, -9V, -14, -18C, -19A, -19F and -23F). The Seropositivity cut-off of the assay was a titer for opsonophagocytic activity higher than or equal to (≥) 8, except for the OPA-19A for which the titer was ≥ to the serotype-specific Lower Limit of Quantification (=143). This outcome concerns results for the Booster Phase of the study.
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 68 | 58 | 68 | 62
Titers
  OPA-1 Month 10: number analyzed (Participants) | 44 | 40 | 45 | 43
  OPA-1 Month 10 | 12.4 [7.6 to 20.1] | 13.2 [8.3 to 21.1] | 18.7 [11.2 to 31.4] | 10.3 [6.8 to 15.5]
  OPA-1 Month 11: number analyzed (Participants) | 68 | 56 | 66 | 59
  OPA-1 Month 11 | 373.5 [253.3 to 550.8] | 369.2 [252.8 to 539.4] | 300.0 [213.2 to 422.1] | 369.3 [281.4 to 484.6]
  OPA-4 Month 10: number analyzed (Participants) | 41 | 36 | 42 | 34
  OPA-4 Month 10 | 36.2 [19.1 to 68.4] | 48.3 [25.6 to 91.0] | 122.3 [75.0 to 199.6] | 18.5 [9.7 to 35.4]
  OPA-4 Month 11: number analyzed (Participants) | 68 | 57 | 68 | 62
  OPA-4 Month 11 | 1370.7 [1034.2 to 1816.6] | 1634.8 [1284.8 to 2080.3] | 2043.3 [1609.1 to 2594.6] | 2882.6 [2252.4 to 3689.1]
  OPA-5 Month 10: number analyzed (Participants) | 44 | 36 | 45 | 42
  OPA-5 Month 10 | 9.3 [6.9 to 12.5] | 10.5 [6.9 to 16.1] | 9.5 [6.9 to 12.9] | 8.7 [6.3 to 12.0]
  OPA-5 Month 11: number analyzed (Participants) | 68 | 56 | 66 | 61
  OPA-5 Month 11 | 154.5 [111.8 to 213.4] | 166.8 [118.4 to 234.8] | 139.3 [102.3 to 189.8] | 327.4 [254.2 to 421.8]
  OPA-6B Month 10: number analyzed (Participants) | 36 | 36 | 40 | 36
  OPA-6B Month 10 | 103.2 [56.5 to 188.4] | 174.5 [102.1 to 298.2] | 136.9 [76.1 to 246.4] | 113.8 [59.3 to 218.6]
  OPA-6B Month 11: number analyzed (Participants) | 66 | 58 | 68 | 62
  OPA-6B Month 11 | 802.1 [531.7 to 1210.0] | 700.3 [481.3 to 1018.8] | 1013.8 [744.6 to 1380.3] | 2731.1 [1972.7 to 3781.1]
  OPA-7F Month 10: number analyzed (Participants) | 42 | 38 | 46 | 40
  OPA-7F Month 10 | 795.5 [560.1 to 1129.9] | 886.4 [599.1 to 1311.5] | 1322.5 [961.5 to 1819.1] | 1895.8 [1420.6 to 2530.0]
  OPA-7F Month 11: number analyzed (Participants) | 68 | 55 | 64 | 61
  OPA-7F Month 11 | 5819.9 [4473.1 to 7572.2] | 5733.8 [4165.0 to 7893.5] | 8336.9 [6357.9 to 10931.8] | 18012.3 [13872.4 to 23387.7]
  OPA-9V Month 10: number analyzed (Participants) | 39 | 37 | 40 | 38
  OPA-9V Month 10 | 281.5 [175.4 to 451.7] | 340.8 [224.0 to 518.5] | 433.7 [318.3 to 591.0] | 510.4 [344.6 to 755.8]
  OPA-9V Month 11: number analyzed (Participants) | 68 | 56 | 67 | 61
  OPA-9V Month 11 | 2001.6 [1506.6 to 2659.3] | 2436.5 [1734.5 to 3422.6] | 3711.7 [2881.2 to 4781.4] | 6839.2 [5464.7 to 8559.3]
  OPA-14 Month 10: number analyzed (Participants) | 35 | 34 | 40 | 32
  OPA-14 Month 10 | 275.8 [175.2 to 434.3] | 208.1 [111.9 to 386.9] | 355.6 [216.3 to 584.8] | 483.0 [286.9 to 813.1]
  OPA-14 Month 11: number analyzed (Participants) | 68 | 55 | 68 | 61
  OPA-14 Month 11 | 2216.9 [1678.0 to 2928.9] | 2297.4 [1640.0 to 3218.4] | 2488.9 [1942.5 to 3189.0] | 3545.0 [2465.2 to 5097.8]
  OPA-18C Month 10: number analyzed (Participants) | 36 | 35 | 35 | 28
  OPA-18C Month 10 | 5.1 [4.0 to 6.6] | 6.3 [4.6 to 8.7] | 6.7 [4.9 to 9.0] | 4.8 [3.9 to 6.1]
  OPA-18C Month 11: number analyzed (Participants) | 68 | 55 | 62 | 60
  OPA-18C Month 11 | 374.6 [271.2 to 517.4] | 303.6 [197.7 to 466.3] | 511.0 [356.7 to 732.2] | 464.4 [327.7 to 658.1]
  OPA-19F Month 10: number analyzed (Participants) | 42 | 40 | 46 | 41
  OPA-19F Month 10 | 18.0 [11.2 to 29.0] | 31.0 [19.2 to 49.9] | 30.7 [19.2 to 49.2] | 7.4 [4.8 to 11.5]
  OPA-19F Month 11: number analyzed (Participants) | 67 | 56 | 66 | 61
  OPA-19F Month 11 | 650.2 [444.1 to 951.9] | 778.9 [500.4 to 1212.3] | 1053.9 [812.6 to 1366.8] | 767.1 [582.1 to 1010.9]
  OPA-23F Month 10: number analyzed (Participants) | 41 | 35 | 42 | 37
  OPA-23F Month 10 | 189.6 [83.5 to 430.5] | 281.4 [123.2 to 642.8] | 242.5 [106.5 to 552.2] | 367.4 [150.3 to 897.8]
  OPA-23F Month 11: number analyzed (Participants) | 68 | 56 | 66 | 60
  OPA-23F Month 11 | 3621.0 [2534.5 to 5173.2] | 2563.6 [1831.6 to 3588.2] | 4465.4 [3368.6 to 5919.3] | 32508.0 [23754.9 to 44486.3]
  OPA-3 Month 10: number analyzed (Participants) | 31 | 23 | 30 | 24
  OPA-3 Month 10 | 6.7 [4.7 to 9.5] | 8.3 [4.9 to 14.0] | 6.3 [4.6 to 8.8] | 12.0 [7.6 to 19.1]
  OPA-3 Month 11: number analyzed (Participants) | 64 | 48 | 65 | 60
  OPA-3 Month 11 | 7.8 [5.7 to 10.6] | 7.8 [5.4 to 11.2] | 9.2 [6.8 to 12.5] | 333.9 [260.3 to 428.3]
  OPA-6A Month 10: number analyzed (Participants) | 41 | 35 | 42 | 35
  OPA-6A Month 10 | 26.5 [13.2 to 52.9] | 23.3 [10.3 to 53.1] | 18.7 [9.8 to 35.7] | 129.7 [61.2 to 274.7]
  OPA-6A Month 11: number analyzed (Participants) | 64 | 57 | 67 | 61
  OPA-6A Month 11 | 163.1 [94.0 to 283.1] | 190.0 [106.6 to 338.4] | 276.2 [174.8 to 436.6] | 4855.3 [3606.3 to 6536.8]
  OPA-19A Month 10: number analyzed (Participants) | 38 | 30 | 34 | 46
  OPA-19A Month 10 | 211.8 [139.2 to 322.4] | 262.0 [157.8 to 435.1] | 315.6 [193.5 to 514.6] | 776.3 [542.2 to 1111.7]
  OPA-19A Month 11: number analyzed (Participants) | 47 | 42 | 53 | 47
  OPA-19A Month 11 | 2006.3 [1539.1 to 2615.3] | 2609.5 [1919.1 to 3548.2] | 2699.1 [2262.2 to 3220.5] | 7137.0 [5909.4 to 8619.6]

12. Secondary Outcome: Concentrations of Antibodies Inhibiting Pneumococcal Pneumolysin Toxoid Haemolysis Activity - Primary Phase of the Study
Description: Analysis of the concentrations of antibodies inhibiting pneumococcal pneumolysin toxoid haemolysis activity (anti-Ply) was not performed as no assay was validated to perform this analysis. This outcome concerns results for the Primary Phase of the study.
Time Frame: At Month 3, e. g. one month post-Dose 3 of pneumococcal vaccine (10PP, Synflorix™ or Prevnar 13™)
Population: This analysis could not be performed as no validated assay was available.
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Concentrations of Antibodies Inhibiting Pneumococcal Pneumolysin Toxoid Haemolysis Activity - Booster Phase of the Study
Description: Analysis of the concentrations of antibodies inhibiting pneumococcal pneumolysin toxoid haemolysis activity (anti-Ply) was not performed as no assay was validated to perform this analysis. This outcome concerns results for the Booster Phase of the study.
Time Frame: as for outcome 5
Population: This analysis could not be performed as no validated assay was available.
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Concentrations of Antibodies Against Diphtheria (Anti-D) and Tetanus (Anti-T) - Primary Phase of the Study
Description: Antibody concentrations will be expressed as geometric mean concentrations (GMCs) in International Units per milliliter (IU/mL). The seroprotection cut-off of the assay was an antibody concentration higher than or equal to (≥) 0.1 IU/mL. This outcome concerns results for the Primary Phase of the study.
Time Frame: At Month 3, e. g. one month post-Dose 3 of pneumococcal vaccine (10PP, Synflorix™ or Prevnar 13™)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 59 | 54 | 57 | 60
IU/mL
  ANTI-D At Month 3 | 3.251 [2.729 to 3.873] | 3.185 [2.556 to 3.968] | 3.353 [2.756 to 4.080] | 2.933 [2.464 to 3.492]
  ANTI-T At Month 3 | 2.579 [2.187 to 3.041] | 2.193 [1.819 to 2.643] | 2.252 [1.930 to 2.627] | 1.416 [1.166 to 1.719]

15. Secondary Outcome: Concentrations of Antibodies Against Diphtheria (Anti-D) and Tetanus (Anti-T) - Booster Phase of the Study
Description: Antibody concentrations will be expressed as geometric mean concentrations (GMCs) in International Units per milliliter (IU/mL). The seroprotection cut-off of the assay was an antibody concentration higher than or equal to (≥) 0.1 IU/mL. This outcome concerns results for the Booster Phase of the study.
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 45 | 50 | 46 | 49
IU/mL
  ANTI-D At Month 10: number analyzed (Participants) | 43 | 50 | 42 | 49
  ANTI-D At Month 10 | 0.731 [0.575 to 0.929] | 0.587 [0.461 to 0.747] | 0.651 [0.507 to 0.836] | 0.614 [0.497 to 0.758]
  ANTI-D At Month 11: number analyzed (Participants) | 45 | 47 | 46 | 48
  ANTI-D At Month 11 | 9.872 [8.191 to 11.898] | 8.688 [7.026 to 10.743] | 9.742 [7.991 to 11.878] | 8.290 [6.943 to 9.899]
  ANTI-T At Month 10: number analyzed (Participants) | 43 | 50 | 42 | 49
  ANTI-T At Month 10 | 0.815 [0.665 to 0.999] | 0.727 [0.570 to 0.927] | 0.726 [0.604 to 0.874] | 0.371 [0.280 to 0.493]
  ANTI-T At Month 11: number analyzed (Participants) | 45 | 47 | 46 | 48
  ANTI-T At Month 11 | 8.725 [7.259 to 10.488] | 8.703 [7.415 to 10.215] | 9.929 [8.653 to 11.394] | 5.040 [4.074 to 6.234]

16. Secondary Outcome: Concentrations of Antibodies Against Pertussis Toxoid (Anti-PT), Filamentous Haemagglutinin (Anti-FHA), Pertactin (Anti-PRN) - Primary Phase of the Study
Description: Antibody concentrations will be measured by enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs) in Elisa Units per milliliter (EL.U/mL). The seropositivity cut-off of the assay was an antibody concentration higher than or equal to (≥) 5 EL.U/mL. This outcome concerns results for the primary Phase of the study.
Time Frame: At Month 3, e. g. one month post-Dose 3 of pneumococcal vaccine (10PP, Synflorix™ or Prevnar 13™)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 59 | 54 | 57 | 60
EL.U/mL
  ANTI-PT At Month 3: number analyzed (Participants) | 59 | 54 | 57 | 59
  ANTI-PT At Month 3 | 69.0 [59.9 to 79.4] | 64.3 [54.8 to 75.3] | 70.0 [61.6 to 79.4] | 64.6 [53.2 to 78.3]
  ANTI-FHA At Month 3 | 187.9 [159.0 to 222.1] | 178.1 [150.2 to 211.2] | 157.1 [132.5 to 186.3] | 188.6 [156.4 to 227.5]
  ANTI-PRN At Month 3 | 95.1 [79.2 to 114.4] | 79.5 [63.6 to 99.2] | 91.4 [75.2 to 111.1] | 87.2 [70.6 to 107.5]

17. Secondary Outcome: Concentrations of Antibodies Against Pertussis Toxoid (Anti-PT), Filamentous Haemagglutinin (Anti-FHA), Pertactin (Anti-PRN) - Booster Phase of the Study
Description: Antibody concentrations will be measured by enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs) in Elisa Units per milliliter (EL.U/mL). The seropositivity cut-off of the assay was an antibody concentration higher than or equal to (≥) 5 EL.U/mL. This outcome concerns results for the Booster Phase of the study.
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 45 | 50 | 46 | 49
EL.U/mL
  ANTI-PT At Month 10: number analyzed (Participants) | 43 | 50 | 42 | 49
  ANTI-PT At Month 10 | 17.5 [13.4 to 22.9] | 12.7 [9.9 to 16.3] | 12.1 [9.7 to 15.1] | 12.2 [9.6 to 15.5]
  ANTI-PT At Month 11: number analyzed (Participants) | 45 | 47 | 46 | 48
  ANTI-PT At Month 11 | 93.8 [75.4 to 116.6] | 90.6 [73.5 to 111.7] | 95.7 [80.1 to 114.3] | 85.2 [70.3 to 103.2]
  ANTI-FHA At Month 10: number analyzed (Participants) | 43 | 50 | 42 | 49
  ANTI-FHA At Month 10 | 63.0 [50.3 to 78.9] | 51.7 [40.1 to 66.6] | 48.5 [38.3 to 61.5] | 54.2 [42.5 to 69.2]
  ANTI-FHA At Month 11: number analyzed (Participants) | 45 | 47 | 46 | 48
  ANTI-FHA At Month 11 | 359.4 [291.3 to 443.5] | 380.1 [311.9 to 463.2] | 308.4 [252.0 to 377.3] | 376.7 [322.6 to 439.8]
  ANTI-PRN At Month 10: number analyzed (Participants) | 43 | 50 | 42 | 49
  ANTI-PRN At Month 10 | 21.8 [15.8 to 30.1] | 16.1 [11.7 to 22.2] | 14.3 [10.7 to 19.3] | 14.3 [10.6 to 19.3]
  ANTI-PRN At Month 11: number analyzed (Participants) | 45 | 47 | 46 | 48
  ANTI-PRN At Month 11 | 294.8 [227.0 to 382.8] | 228.5 [174.2 to 299.7] | 224.2 [180.0 to 279.1] | 197.3 [154.3 to 252.2]

18. Secondary Outcome: Concentrations of Antibodies Against Hepatitis B (Anti-HBs) - Primary Phase of the Study
Description: Antibody concentrations will be expressed as geometric mean concentrations (GMCs) in milli-International Units per milliliter (mIU/mL). The seroprotection cut-off of the assay was an antibody concentration higher than or equal to (≥) 10 mIU/mL. This outcome concerns results for the Primary Phase of the study. Note that the percentage of subjects with concentration ≥10 mIU/mL was over-estimated due to the use of in-house assay overestimating concentrations between 10-100 mIU/mL. Accordingly GMCs were also overestimated.
Time Frame: At Month 3, e. g. one month post-Dose 3 of pneumococcal vaccine (10PP, Synflorix™ or Prevnar 13™)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 50 | 43 | 47 | 48
mIU/mL | 676.7 [466.2 to 982.3] | 619.1 [386.5 to 991.5] | 719.8 [537.0 to 965.0] | 877.4 [597.0 to 1289.4]

19. Secondary Outcome: Concentrations of Antibodies Against Hepatitis B (Anti-HBs) - Booster Phase of the Study
Description: Antibody concentrations will be expressed as geometric mean concentrations (GMCs) in milli-International Units per milliliter (mIU/mL). The seroprotection cut-off of the assay was an antibody concentration higher than or equal to (≥) 10 mIU/mL. This outcome concerns results for the Booster Phase of the study. * A decrease in the specificity of the anti-HB Enzyme-Linked ImmunoSorbent Assay (ELISA) assay had been observed in some studies for low levels of antibody (10-100 mIU/mL). The table shows updated results following partial or complete reanalysis. The retest has been performed in using Food and Drug Administration (FDA)-approved ChemiLuminescence ImmunoAssay (CLIA) commercial assay Centaur™.
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 60 | 65 | 62 | 64
mIU/mL
  ANTI-HBs At Month 10: number analyzed (Participants) | 50 | 46 | 47 | 54
  ANTI-HBs At Month 10 | 299.2 [199.0 to 449.8] | 287.1 [195.1 to 422.4] | 166.6 [105.2 to 263.8] | 174.5 [113.5 to 268.2]
  ANTI-HBs At Month 11 | 4110.9 [2576.5 to 6558.9] | 4234.8 [2961.4 to 6055.7] | 3142.4 [2151.1 to 4590.6] | 3116.4 [2142.5 to 4533.0]

20. Secondary Outcome: Concentrations of Antibodies Against Polyribosyl Ribitol Phosphate (Anti-PRP) - Primary Phase of the Study
Description: Antibody concentrations will be expressed as geometric mean concentrations (GMCs) in microgram per milliliter (µg/mL). The seroprotection cut-off of the assay was an antibody concentration higher than or equal to (≥) 0.15 µg/mL or 1 µg/mL. This outcome concerns results for the Primary Phase of the study.
Time Frame: At Month 3, e. g. one month post-Dose 3 of pneumococcal vaccine (10PP, Synflorix™ or Prevnar 13™)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 59 | 54 | 57 | 60
µg/mL | 1.920 [1.433 to 2.573] | 1.975 [1.390 to 2.806] | 1.813 [1.330 to 2.472] | 0.963 [0.690 to 1.344]

21. Secondary Outcome: Concentrations of Antibodies Against Polyribosyl Ribitol Phosphate (Anti-PRP) - Booster Phase of the Study
Description: Antibody concentrations will be expressed as geometric mean concentrations (GMCs) in microgram per milliliter (µg/mL). The seroprotection cut-off of the assay was an antibody concentration higher than or equal to (≥) 0.15 µg/mL or 1 µg/mL. This outcome concerns results for the Booster Phase of the study.
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 45 | 50 | 46 | 49
µg/mL
  ANTI-PRP At Month 10: number analyzed (Participants) | 43 | 50 | 42 | 49
  ANTI-PRP At Month 10 | 0.390 [0.279 to 0.546] | 0.446 [0.306 to 0.651] | 0.503 [0.360 to 0.703] | 0.272 [0.193 to 0.384]
  ANTI-PRP At Month 11: number analyzed (Participants) | 45 | 47 | 46 | 48
  ANTI-PRP At Month 11 | 16.961 [11.652 to 24.689] | 28.168 [20.580 to 38.554] | 24.549 [16.379 to 36.795] | 12.853 [8.301 to 19.899]

22. Secondary Outcome: Titers of Antibodies Against Poliovirus Types 1, 2 and 3 (Anti-1, Anti-2 and Anti-3) - Primary Phase of the Study
Description: Antibody titers will be measured by virus microneutralization test, expressed as geometric mean titers (GMTs). The cut-off of the assay for anti-1, anti-2 and anti-3 antibody was a titer higher than or equal to (≥) 8. This outcome concerns results for the Primary Phase of the study.
Time Frame: At Month 3, e. g. one month post-Dose 3 of pneumococcal vaccine (10PP, Synflorix™ or Prevnar 13™)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 45 | 37 | 43 | 42
Titers
  ANTI-Polio 1 At Month 3: number analyzed (Participants) | 45 | 37 | 43 | 41
  ANTI-Polio 1 At Month 3 | 175.7 [124.5 to 247.8] | 138.2 [91.0 to 209.8] | 190.3 [115.7 to 312.9] | 173.7 [128.9 to 234.0]
  ANTI-Polio 2 At Month 3: number analyzed (Participants) | 44 | 28 | 36 | 42
  ANTI-Polio 2 At Month 3 | 134.3 [86.3 to 209.1] | 114.7 [68.6 to 192.0] | 177.6 [102.5 to 307.8] | 148.4 [101.1 to 217.9]
  ANTI-Polio 3 At Month 3: number analyzed (Participants) | 45 | 37 | 41 | 41
  ANTI-Polio 3 At Month 3 | 445.7 [290.9 to 682.9] | 432.2 [273.0 to 684.3] | 552.7 [361.1 to 846.1] | 538.6 [413.6 to 701.4]

23. Secondary Outcome: Titers of Antibodies Against Poliovirus Types 1, 2 and 3 (Anti-1, Anti-2 and Anti-3) - Booster Phase of the Study
Description: Antibody titers will be measured by virus microneutralization test, expressed as geometric mean titers (GMTs). The cut-off of the assay for anti-1, anti-2 and anti-3 antibody was a titer higher than or equal to (≥) 8. This outcome concerns results for the Booster Phase of the study.
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 42 | 46 | 36 | 43
Titers
  ANTI-Polio 1 At Month 10: number analyzed (Participants) | 35 | 37 | 32 | 41
  ANTI-Polio 1 At Month 10 | 41.7 [25.9 to 67.3] | 58.3 [35.6 to 95.6] | 55.5 [33.9 to 90.9] | 55.4 [38.3 to 80.1]
  ANTI-Polio 1 At Month 11: number analyzed (Participants) | 40 | 41 | 30 | 41
  ANTI-Polio 1 At Month 11 | 1116.0 [696.1 to 1789.3] | 1222.0 [737.1 to 2026.1] | 1149.6 [764.3 to 1729.0] | 1233.2 [898.9 to 1691.9]
  ANTI-Polio 2 At Month 10: number analyzed (Participants) | 39 | 46 | 36 | 43
  ANTI-Polio 2 At Month 10 | 50.4 [33.4 to 76.0] | 55.9 [35.6 to 87.8] | 61.0 [40.2 to 92.7] | 66.8 [48.6 to 91.9]
  ANTI-Polio 2 At Month 11: number analyzed (Participants) | 42 | 40 | 34 | 38
  ANTI-Polio 2 At Month 11 | 1998.1 [1415.0 to 2821.5] | 2332.2 [1739.0 to 3127.6] | 2048.3 [1484.6 to 2825.9] | 2284.8 [1705.1 to 3061.6]
  ANTI-Polio 3 At Month 10: number analyzed (Participants) | 36 | 40 | 33 | 38
  ANTI-Polio 3 At Month 10 | 167.7 [113.3 to 248.3] | 104.9 [68.7 to 160.2] | 125.4 [81.2 to 193.6] | 93.1 [66.2 to 130.9]
  ANTI-Polio 3 At Month 11: number analyzed (Participants) | 41 | 37 | 34 | 39
  ANTI-Polio 3 At Month 11 | 2995.8 [2081.1 to 4312.6] | 3626.3 [2623.6 to 5012.2] | 2696.8 [1913.7 to 3800.4] | 2820.0 [2127.9 to 3737.4]

24. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms - Primary Phase of the Study
Description: Assessed local symptoms were pain, redness and swelling at injection site. Any = Occurrence of the specified solicited local symptom, regardless of intensity. Grade 3 Pain = Crying when limb was moved/spontaneously painful. Grade 3 Redness/Swelling = Redness/swelling at injection site larger than (>) 30 millimeters (mm).
Time Frame: Within the 7-day (Days 0-6) periods post vaccination, after each dose (D) of the 3-dose primary vaccination course
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 146 | 142 | 144 | 142
Participants
  Any Pain, post D1 | 52 | 46 | 53 | 40
  Grade 3 Pain, post D1 | 0 | 2 | 3 | 0
  Any Redness, post D1 | 59 | 58 | 52 | 51
  Grade 3 Redness, post D1 | 0 | 0 | 3 | 2
  Any Swelling, post D1 | 47 | 46 | 34 | 37
  Grade 3 Swelling, post D1 | 3 | 5 | 3 | 6
  Any Pain, post D2 | 52 | 49 | 42 | 43
  Grade 3 Pain, post D2 | 2 | 0 | 1 | 2
  Any Redness, post D2 | 67 | 67 | 63 | 59
  Grade 3 Redness, post D2 | 2 | 2 | 3 | 0
  Any Swelling, post D2 | 49 | 56 | 43 | 38
  Grade 3 Swelling, post D2 | 5 | 4 | 2 | 3
  Any Pain, post D3: number analyzed (Participants) | 146 | 141 | 143 | 142
  Any Pain, post D3 | 41 | 35 | 37 | 45
  Grade 3 Pain, post D3: number analyzed (Participants) | 146 | 141 | 143 | 142
  Grade 3 Pain, post D3 | 2 | 3 | 1 | 1
  Any Redness, post D3: number analyzed (Participants) | 146 | 141 | 143 | 142
  Any Redness, post D3 | 65 | 65 | 58 | 65
  Grade 3 Redness, post D3: number analyzed (Participants) | 146 | 141 | 143 | 142
  Grade 3 Redness, post D3 | 3 | 2 | 0 | 3
  Any Swelling, post D3: number analyzed (Participants) | 146 | 141 | 143 | 142
  Any Swelling, post D3 | 52 | 52 | 43 | 43
  Grade 3 Swelling, post D3: number analyzed (Participants) | 146 | 141 | 143 | 142
  Grade 3 Swelling, post D3 | 6 | 3 | 3 | 5

25. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms - Booster Phase of the Study
Description: as for outcome 24
Time Frame: Within the 7-day (Days 0-6) period after booster vaccination
Population: The analysis was performed on the Total Vaccinated cohort for the Booster Phase, which included all subjects who received the booster dose of vaccine against pneumococcal diseases, with analysis done solely on subjects with post-vaccination solicited symptoms results available.
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 144 | 140 | 139 | 140
Participants
  Any Pain | 77 | 73 | 61 | 68
  Grade 3 Pain | 7 | 6 | 3 | 4
  Any Redness | 83 | 81 | 68 | 66
  Grade 3 Redness | 11 | 15 | 12 | 7
  Any Swelling | 70 | 55 | 49 | 59
  Grade 3 Swelling | 8 | 8 | 7 | 10

26. Secondary Outcome: Number of Subjects With Any, Grade 3 Solicited General Symptoms and Solicited General Symptoms With Relationship to Vaccination - Booster Phase of the Study
Description: Assessed solicited general symptoms were Drowsiness, Irritability, Loss of appetite (Loss Appet.) and Fever (rectal temperature higher than [≥] 38 degrees Celsius [°C]). Any = Occurrence of the specified solicited general symptom, regardless of intensity and relationship to vaccination. Related = Occurrence of the specified symptom assessed by the investigator as causally related to vaccination. Grade 3 Drowsiness = Drowsiness that prevented normal activity. Grade 3 Irritability = Crying that could not be comforted/prevented normal activity. Grade 3 Loss of appetite = Subject did not eat at all. Grade 3 Fever = Axillary temperature higher than (>) 40.0°C.
Time Frame: Within the 7-day (Days 0-6) period post vaccination after booster vaccination
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 144 | 140 | 139 | 140
Participants
  Any Drowsiness | 77 | 64 | 66 | 73
  Grade 3 Drowsiness | 1 | 5 | 1 | 1
  Related Drowsiness | 68 | 61 | 59 | 69
  Any Irritability | 95 | 84 | 82 | 90
  Grade 3 Irritability | 12 | 8 | 4 | 8
  Related Irritability | 86 | 82 | 76 | 83
  Any Loss Appet | 49 | 38 | 36 | 57
  Grade 3 Loss Appet. | 3 | 4 | 2 | 2
  Related Loss Appet. | 42 | 38 | 33 | 49
  Any Fever | 50 | 55 | 51 | 53
  Grade 3 Fever | 1 | 0 | 1 | 3
  Related Fever | 44 | 52 | 45 | 47

27. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs) - Primary Phase of the Study
Description: An unsolicited AE was defined as any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For the marketed products administered in the study, this also included failure to produce expected benefits (i.e. lack of efficacy), abuse or misuse of the product. Any = Occurrence of an unsolicited AE, regardless of intensity or relationship to vaccination.
Time Frame: Within the 31-day (Days 0-30) period post primary vaccination, across doses
Population: The analysis was performed on the Total Vaccinated cohort for the Primary Phase, which included all vaccinated subjects with at least one of the 3 vaccine doses against pneumococcal diseases.
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 146 | 142 | 145 | 142
Participants | 55 | 68 | 64 | 61

28. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs) - Booster Phase of the Study
Description: as for outcome 27
Time Frame: Within the 31-day (Days 0-30) period post booster vaccination
Population: The analysis was performed on the Total Vaccinated cohort of Booster Phase, which included all subjects who received the booster dose of vaccine against pneumococcal diseases.
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 144 | 140 | 140 | 140
Participants | 40 | 26 | 27 | 34

29. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: An SAE was defined as any medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity in a subject. AE(s) considered as SAE(s) also included invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that did not result in hospitalization, as per the medical or scientific judgement of the physician. Any = Occurrence of an SAE, regardless of relationship to vaccination.
Time Frame: During the entire study period (Months 0-11)
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
Number analyzed (Participants) | 146 | 142 | 145 | 142
Participants | 13 | 9 | 21 | 17

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during the 7 days post-primary vaccination and post-booster vaccination. Unsolicited AEs during 31 days post-primary vaccination and post booster vaccination. SAEs: during the entire study period (Months 0-11).
Description: Solicited symptoms results are presented only for subjects for whom results were available.
Arm/Group | 10PP-LD/Infanrix Hexa Group | 10PP-HD/Infanrix Hexa Group | Synflorix/Infanrix Hexa Group | Prevnar 13/Infanrix Hexa Group
All-Cause Mortality (participants affected / at risk) | 0/146 | 0/142 | 0/145 | 0/142
Serious Adverse Events (participants affected / at risk) | 13/146 | 9/142 | 21/145 | 17/142
Other Adverse Events (participants affected / at risk) | 141/146 | 137/142 | 139/145 | 134/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10PP-LD/Infanrix Hexa Group (N=146) | 10PP-HD/Infanrix Hexa Group (N=142) | Synflorix/Infanrix Hexa Group (N=145) | Prevnar 13/Infanrix Hexa Group (N=142)
Bronchitis (Infections and infestations) | 1 | 1 | 2 | 3
Otitis media (Infections and infestations) | 3 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 1 | 1 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 2
Thermal burn (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 1 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 1
Psychomotor retardation (Psychiatric disorders) | 1 | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Accidental exposure to product by child (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Breath holding (Psychiatric disorders) | 0 | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 1 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0
Exanthema subitum (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Gastroenteritis Escherichia coli (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hypotonia (Nervous system disorders) | 1 | 0 | 0 | 0
Hypotonic-hyporesponsive episode (Nervous system disorders) | 0 | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Rectal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 10PP-LD/Infanrix Hexa Group (N=146) | 10PP-HD/Infanrix Hexa Group (N=142) | Synflorix/Infanrix Hexa Group (N=145) | Prevnar 13/Infanrix Hexa Group (N=142)
Pain (General disorders) | 75 | 73 | 72/144 | 64 — Symptom reported during the 7-day post-primary vaccination periods, across doses
Redness (General disorders) | 96 | 97 | 88/144 | 83 — Symptom reported during the 7-day post-primary vaccination periods, across doses
Swelling (General disorders) | 82 | 74 | 60/144 | 59 — Symptom reported during the 7-day post-primary vaccination periods , across doses
Drowsiness (General disorders) | 107 | 96 | 98/144 | 102 — Symptom reported during the 7-day post-primary vaccination periods, across doses
Irritability (General disorders) | 118 | 113 | 110/144 | 113 — Symptom reported during the 7-day post-primary vaccination periods, across doses
Loss of appetite (General disorders) | 65 | 59 | 59/144 | 57 — Symptom reported during the 7-day post-primary vaccination periods, across doses
Fever (rectal temperature >= 38°C) (General disorders) | 76 | 71 | 74/144 | 65 — Symptom reported during the 7-day post-primary vaccination periods, across doses
Pain (General disorders) | 77/144 | 73/140 | 61/139 | 68/140 — Symptom reported during the 7-day post-booster vaccination period
Redness (General disorders) | 83/144 | 81/140 | 68/139 | 66/140 — Symptom reported during the 7-day post-booster vaccination period
Swelling (General disorders) | 70/144 | 55/140 | 49/139 | 59/140 — Symptom reported during the 7-day post-booster vaccination period
Drowsiness (General disorders) | 77/144 | 64/140 | 66/139 | 73/140 — Symptom reported during the 7-day post-booster vaccination period
Irritability (General disorders) | 95/144 | 84/140 | 82/139 | 90/140 — Symptom reported during the 7-day post-booster vaccination period
Loss of appetite (General disorders) | 49/144 | 38/140 | 36/139 | 57/140 — Symptom reported during the 7-day post-booster vaccination period
Fever (rectal temperature >= 38°C) (General disorders) | 50/144 | 55/140 | 51/139 | 53/140 — Symptom reported during the 7-day post-booster vaccination period
Conjunctivitis (Eye disorders) | 5 | 9 | 5 | 3 — Unsolicited AE reported during the 31-day post-primary vaccination periods, across doses
Bronchitis (Infections and infestations) | 6 | 12 | 11 | 13 — Unsolicited AE reported during the 31-day post-primary vaccination periods, across doses
Nasopharyngitis (Infections and infestations) | 10 | 7 | 12 | 8 — Unsolicited AE reported during the 31-day post-primary vaccination periods, across doses
Nasopharyngitis (Infections and infestations) | 9/144 | 4/140 | 3/140 | 6/140 — Unsolicited AE reported during the 31-day post-booster vaccination period
Rhinitis (Infections and infestations) | 11 | 11 | 12 | 14 — Unsolicited AE reported during the 31-day post-primary vaccination periods, across doses
Viral infection (Infections and infestations) | 0 | 9 | 5 | 3 — Unsolicited AE reported during the 31-day post-primary vaccination periods, across doses

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.